CLINICAL TRIAL: NCT06279325
Title: Analysis of the Effectiveness of a Computerized Cognitive Stimulation Program Designed from Occupational Therapy According to the Level of Cognitive Reserve in Older Adults in Primary Care: Stratified Randomized Clinical Trial Protocol
Brief Title: Effects of a Computerized Cognitive Stimulation Intervention Adapted to the Level of Cognitive Reserve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Estela Calatayud, PhD program in Health Sciences, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C.I. PI23/637
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Stimulation program (Experimental)
  Interventions: Behavioral: Computerized cognitive stimulation program
- Control Group (Active Comparator)
  Interventions: Behavioral: Face-to-face training-explanatory session

INTERVENTIONS:
Behavioral: Computerized cognitive stimulation program — * The cognitive stimulation (CS) program, for the IG, will be previously designed by 2 Occupational Therapy (OT) of the team, and adapted to the computerized format through a platform specialized in cognitive neurorehabilitation. The activities will be designed under OT models: human occupation model and cognitive-perceptual model, so that the different professions, interests and roles are represented, and allow to express different levels of complexity, according to the level of Cognitive Reserve (CR).
  * The cognitive aspects to be worked on are: memory, orientation, language, praxis, gnosis, calculation, perception, logical reasoning, attention-concentration and executive functions.
  * In addition, reinforcement, EF, episodic memory, attention and information processing speed activities will be designed, also according to the CR level.
  Arms: Cognitive Stimulation program
Behavioral: Face-to-face training-explanatory session — The CG will undergo a group and face-to-face training-explanatory session, where the importance of maintaining the usual level of cognitive activity will be emphasized.
  Arms: Control Group

SUMMARY:
Normal ageing presents subtle cognitive changes that can be detected before meeting the criteria for Mild cognitive impairment (MCI). Older people with low cognitive reserve and who receive limited cognitive stimulation are at greater risk of deterioration. In this regard, cognitive stimulation (CS) has been identified as an intervention that reduces this risk, provided that its design considers the differences in the level of cognitive reserve (CR) acquired throughout life and the baseline level of cognitive functioning. The general objective of this study is to evaluate, through a randomized clinical trial, the effectiveness of a computerized cognitive stimulation program, designed and adapted from Occupational Therapy based on the level of cognitive reserve in older adults in Primary Care. 100 participants will be randomized in a stratified manner according to the level of cognitive reserve (high/low), assigning 50 participants to the control group and 50 participants to the intervention group. The intervention group will carry out a computerized cognitive stimulation intervention designed and adapted from occupational therapy according to the level of cognitive reserve, through the "stimulus" platform. The main result expected to be achieved is the improvement of higher brain functions. As secondary results, the investigators expect that those cognitive aspects most vulnerable to ageing will decrease more slowly (in areas such as memory, executive function, attention and processing speed) and that the cognitive reserve of the participants will increase, in addition to being able to balance gender differences in these aspects. The investigators think that these results can positively impact the creation of adapted, meaningful and stimulating CS programs in older adults to prevent MCI and experience healthier ageing.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 60 years.
* With score in Lobo's Mini-cognitive Examination (MEC-35) (Lobo, A., Escolar, V., Ezquerra, J., & Seva Díaz, 1979) between: 28-35 points (Friedman et al., 2012; Vinyoles Bargalló et al., 2002).
* Non-institutionalized persons, belonging to the health centers where the study was conducted.
* With a minimum educational level (knowing how to read and write).
* Who do not present hearing, visual or communication difficulties that would prevent them from completing the cognitive training.

Exclusion Criteria:

* People with mild cognitive impairment or Alzheimer's disease (AD).
* People with significant functional impairment.
* People who have received any type of professionalized cognitive stimulation therapy in the last year.
* People with significant psychiatric conditions, such as major depressive disorder or schizophrenia.
* People who are taking medications that may adversely affect cognitive function, such as anticholinergics, tranquilizers and anticonvulsants.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
MEC-35 (Spanish version of Folstein's Mini-Mental) | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  The primary outcome variable is MEC-35 (Spanish version of Folstein's Mini-Mental): the most widely used cognitive test in Primary Care, adapted by Lobo to the Spanish population (Lobo, A., et al 1979). It evaluates 8 components: temporal orientation, spatial orientation, fixation memory, attention, calculation, short-term memory, language and praxis. Its sensitivity is 85-90% and its specificity 69% (Lobo, A. et al 1999). Although its cut-off point for detecting cognitive impairment is 24, in NC, scores between 28-35 points are considered (Friedman et al., 2012; Vinyoles Bargalló et al., 2002).
Cognitive Reserve Questionnaire (CRQ) | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  To determine the level of cognitive reserve (Landenberger et al., 2019) the most suitable questionnaire is the Cognitive Reserve Questionnaire (CRQ) (Rami et al., 2011). It has eight items with between three and six response options. Each item relieves a CR factor: schooling, parental schooling, courses, occupation, musical training, languages, reading and intellectual games. The maximum score is 25 points. Between 7 and 9 points is considered a medium-low range of CR. Between 10-14 points medium-high range, and ≥15 points, high CR. It is an instrument with high reliability and acceptable convergent validity (Martino et al., 2021).

SECONDARY OUTCOMES:
Set-Test | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  -Set-Test (Pascual, L., Martinez, J., Modrego, P., Mostacero, E., Lopez del Val, J., & Morales, 1990): measures verbal fluency of categorical type: colors, animals, fruits and cities, asking the patient to say elements of the 4 categories in one minute. It presents a sensitivity of 87% and a specificity of 67%.
The SDMT or Symbols and Digits Test | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  The SDMT or Symbols and Digits Test measures EF, processing speed and attention. It is a test with good accuracy, sensitivity and specificity, useful for predicting future MCI. The SDMT card consists of a header with a key that relates the numbers from 1 to 9 with different symbols; the participant has 90 seconds to match a specific number with a particular geometric figure. The response can be written or verbal, and the maximum total response time is five minutes. The ideal cut-off point is 44 points, although 38 points can be used for a more specific result (Baudouin et al., 2009).
Color Word Stroop Test (CWST) | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  Color Word Stroop Test (CWST) (Cheng et al., 2012) assesses perseveration, cognitive flexibility, EF and attention (Uttl & Graf, 1997). It consists of naming a color with and without the presence of conflicting or incongruent stimuli. The test consists of three sheets: in the first one, colors written in black ink are repeated, in the second one colors with their geometric figure, and in the third one colors written in different ink. The correct answers in the three sheets are collected. This test shows a decrease by age and gender (the most impaired EF in men) (Periáñez et al., 2021; Van der Elst et al., 2008). The limits considered normal are 35-65 points (Graf et al., 1995).
Verbal Learning Test (TAVEC) | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  Verbal Learning Test (TAVEC) Spanish version of the California Verbal Learning Test (CVLT). It evaluates learning and episodic memory capacity. The test consists of memorizing a list of 16 words (list A), belonging to four semantic categories, and their subsequent recall. Five trials are repeated and a second list of 16 words (list B) is administered. Subsequently, recall of list A and recall by semantic categories is requested. After about 20 minutes, free recall of word list A and recall by semantic categories is requested again. Both Spearman's coefficient and Cronbach's α indicate high reliability (Nieto Barco et al., 2014).
Mobile Device Proficiency Questionnaire in Short Form (MDPQ-16) | An initial evaluation (pre), post-intervention (in a period of 2 to 7 days after the last intervention session) and two follow-up evaluations (at 6 and 12 months) will be carried out.
  Mobile Device Proficiency Questionnaire in Short Form (MDPQ-16). Tests experience and aptitude for using mobile devices in eight domains: mobile device basics, communication, data and file storage, Internet, calendar, entertainment, privacy, troubleshooting, and software management. Each of the domains is scored on a 5-point scale (e.g., 1 = never tried , 2 = not at all , 3 = not very easily , 4 = somewhat easily , 5 = very easily). The total score ranges from 8 to 40, with higher scores reflecting greater competence. Internal consistency is excellent (Cronbach's α=.96).(Roque & Boot, 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Arrabal, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
The primary objective of this plan is to disseminate individual participant data (IPD) from our research study to a wide audience of researchers and stakeholders. By publishing in open-access journals and presenting at conferences, the investigators aim to maximize the visibility and accessibility of our data, fostering collaboration and advancing scientific knowledge in our field.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Calatayud E, Olivan-Blazquez B, Aguilar-Latorre A, Cuenca-Zaldivar JN, Magallon-Botaya RM, Gomez-Soria I. Digital Competence and Cognitive Reserve in Relation to Different Domains of Cognitive Functioning in Older Adults and Factors Modulating This Association: A Cross-Sectional Study of a Randomized Clinical Trial. Geriatr Gerontol Int. 2025 Nov;25(11):1525-1535. doi: 10.1111/ggi.70199. Epub 2025 Oct 8. PMID 41060253